CLINICAL TRIAL: NCT00885560
Title: Do People With ADHD, Who Respond Well to Amphetamine Medication But Not to Methylphenidate, Have Allelic Variants of the SNAP 25 Gene?
Brief Title: SNAP 25 Gene Study
Status: Terminated | Type: Observational
Why Stopped: Collecting data for the population involved was very difficult. Over 3 years, only 19 participants were recruited.
Sponsor: University of British Columbia (Other)
Collaborators: UBC Human Early Learning Partnership (HELP) (Unknown)
Responsible Party: Sponsor
Other Study IDs: H05-70410
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: ADHD; SNAP 25; amphetamine; methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood for genetic analysis.
Oversight: Data Monitoring Committee: No

SUMMARY:
To enhance our capacity to correctly choose the appropriate medication for ADHD patients on the first try based on the presence of a particular variant of a gene that could be identified on a laboratory test. It is hypothesized that patients with Attention Deficit Hyperactivity Disorder (ADHD) who have failed to respond to methylphenidate medication, but do respond to amphetamines, have a higher than expected incidence the allelic variants of the SNAP 25 gene associated with ADHD, and mutations of the dopamine system genes DRD1, 2, 4, 5 and dopamine transporter and COMTand MAOA.

DETAILED DESCRIPTION:
Previous research has demonstrated that while 75% of patients respond to any stimulant, of those who do not 33% will respond to a stimulant of the other class. Based on previous research correlating increased mutations in the dopamine system genes DRD1, 2, 4, 5, dopamine transporter, COMT, and MAOA with ADHD, we will also be investigating the relationship between mutations in these genes and patient response to MPH and amphetamines. This study is a pilot, but it was an obvious next step in the studies that are being done on the genetics of ADHD. The outcome of this research, whether an association is or is not found, will be of considerable interest to researchers internationally, and will demonstrate the value of HELP funding in promoting research that can alleviate mental illness in children The study will make a significant contribution to appropriate intervention for these children, and promote greater awareness that the deficits suffered by children with attention problems is neither willful nor a matter of intelligence, but rather a syndrome that can be explained and can be modified with appropriate medical care.

A chi-square test will be conducted to determine whether there is differential representation of SNAP 25 among therapeutic methylphenidate responders versus non-responders. Statistical comparison will be performed using a two-tailed test at the .05 level of significance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be male or female outpatients who are at least 6 years of age (there is no upper age limit)
2. Patients must meet DSM-IV criteria for ADHD
3. Patients and parents/guardians must have a degree of understanding sufficient to be able to communicate suitably with the investigator and study coordinator
4. Patients must have tolerated the drug at therapeutic doses, but have shown a true lack of improvement in symptoms
5. Must have shown clinically significant superiority in improvement in ADHD symptoms on amphetamine relative to MPH.

Exclusion Criteria:

1. Must not have a true allergy to methylphenidate or amphetamines
2. Must not have a history of serious adverse reactions to methylphenidate

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: ADHD patients from 6 years of age
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2006-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret D. Weiss, MD, Ph.D, Principal Investigator — University of British Columbia; Jim Kennedy, MD, Study Director — University of British Columbia; Atilla Turgay, MD, Study Director — British Columbia Children's & Women's Hospital
Locations (1):
- Provincial ADHD Program, BC Children's & Women's Health Centre, Vancouver, British Columbia, Canada